CLINICAL TRIAL: NCT02174107
Title: Health Economics Evaluation of Percutaneous Vertebroplasty Compared to Radiation Therapy in Patients With Painful Spine Metastases.
Acronym: Radiointer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment issues due to feasability issues in centers
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RADIOINTER01
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Spine Metastases
Keywords: Health economics; Percutaneous vertebroplasty; Radiation therapy; Painful spine metastases
MeSH Terms: interventions — Vertebroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Percutaneous vertebroplasty
  Interventions: Procedure: Percutaneous vertebroplasty
- Arm B (Experimental): External radiotherapy
  Interventions: Radiation: External radiotherapy

INTERVENTIONS:
Radiation: External radiotherapy — The radiation technique used for each patient will be based on local clinical practices and on number of vertebae to treat between 1*8 Gy; 5*4 Gy and 10*3 Gy
  Arms: Arm B
Procedure: Percutaneous vertebroplasty
  Other Names: Vertebroplasty
  Arms: Arm A

SUMMARY:
The purpose of this study is to evaluate cost-utility analysis in order to provide recommendations to French decision-makers between vertebroplasty and radiation therapy in Bone spine metastases. Indeed, radiation therapy is often advocated a systematic way. The object of this study would be to expand the use of vertebroplasty.

Moreover, this study assess to the strategy impact on the pain control reduction and functional preservation. In fact, analgesic effect is achieved differently depending on the procedure used.Eligible patients will be recruited and registered consecutively. Patients will be randomly,

This is a health-economic multicenter, prospective, randomized with stratification according to number of vertebrae to treat (1-3 vertebrae vs 4-6 vertebrae) and center :

* Arm A: Percutaneous vertebroplasty
* Arm B: External radiotherapy

This is an open-label study. The expected total study period is 2.5 years (enrolment: 2 years, patient follow-up: 6 months). A total number of 304 patients with spine metastases will be recruited (152 patients/arm).

DETAILED DESCRIPTION:
Bone is the most common site for metastasis. In breast and prostate cancers, 70% of patients dying of their cancer have evidence of metastatic bone disease [Coleman, 2006]. Depending on their localization, bone metastases can have debilitating consequences resulting in considerable morbidity and complex demands on health care resources. Bone spine metastases are the most frequent site observed in patients with cancer of the lung, prostate, breast and hemopoetic organs. The occurrence of spinal metastases in patients with advanced cancer can cause significant morbidity, with pain and/or neurological deficit adversely affecting the patients' quality of life.

Interventional radiology takes a large place in the treatment of bone metastases. Currently, vertebroplasty appears as the most satisfactory technique for stabilization of spine metastases offering a significant improvement of the quality of life. The analgesic effect is achieved very rapidly, i.e. usually within 24 hours post-procedure. Based on several publications, around 90% of patients reported rapid pain relief following vertebroplasty with 60 to 70% of complete pain relief [Mendel, 2009].

Radiotherapy also plays a very important role in the palliative treatment of the metastatic bone. Radiotherapy is effective and well tolerated. A reduction of the pain is noticed for 70 to 80 % of the patients and begins one or two weeks after the treatment. In all, the radiotherapy increases the quality of life of the patients and can reduce the intake of analgesics [Lutz, 2011].

In a lot of cases, vertebroplasty or radiotherapy can both be performed for a same painful patient (the National Institute for Health and Clinical Excellence (NICE) approved the use of vertebroplasty for patients with spinal metastases in November 2008). Radiotherapy remains the gold-standard treatment. However, vertebroplasty could be less costly and more effective compare to radiotherapy. In fact, the superiority of vertebroplasty has been demonstrated at least in the acute post-therapeutic period with (i) more rapid autonomy recovery, (ii) reduction of antalgic intakes, and potentially less side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the day of consenting to the study
* Patient with at least a painful spine metastasis confirmed by MRI / CT scan,
* Localized pain at the lesion ≥ 4 (VAS),
* Bone axial metastasis localised on ≤ 6 different vertebrae,
* Histologically established diagnosis of cancer (lung, kidney, breast, prostate, melanoma, soft tissue sarcomas) other than hematologic malignancy, myeloma, brain tumor, germ cell tumor and bone sarcomas
* ECOG performance status 0 to 2 (Appendix 2)
* Minimum life expectancy of 6 months (Tokuhashi score > 8 )
* Ability to understand and willingness for follow-up visits.
* Covered by a medical insurance
* Signed and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrolment

Exclusion Criteria:

* Solitary metastasis
* SBRT indication
* Contra-indication to vertebroplasty
* Previous radiotherapy for pain management in the same area.
* Patient unable to lie prone
* Neurological deficit due to spinal cord compression,
* Active infection,
* Bleeding risk (platelets < 50000 and PTT > 1.5*ULN),
* Risk of vertebral collapse (SINS score ≥ 13),
* Impossible follow-up for social, geographical, familial or psychological reasons,
* Patient deprived of freedom,
* Patient enrolled in another experimental surgical trial, with therapeutic endpoint,
* Pregnant or breastfeeding women,Pregnant or breastfeeding women (mandatory negative serum or urinary pregnancy test at study entry for all women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Health economics evaluation | 6 months after the end ot treatment
  To perform a cost-utility analysis in order to provide recommendations to French decision-makers on the treatment of patients with painful spine metastases.
  Incremental cost-effectiveness ratio expressed in cost per quality adjusted life year (QALY) gained

SECONDARY OUTCOMES:
Budget impact analysis of vertebroplasty | 6 months after the end of treatment
  Cost-assessment, Quality of life (EQ-5D) Quality adjusted life year,

OTHER OUTCOMES:
Assessment of pain reduction | 3 weeks, 3 months and 6 months after the end of treatment
  Visual analogue scale: VAS

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand BR RICHIOUD, MD, Principal Investigator — Center Leon Berard
Locations (7):
- France (7):
  - Institut Bergonié, Bordeaux
  - Centre Leon Berard, Lyon
  - HCL- Hopital Edouard Herriot, Lyon
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Centre Paul Strauss, Strasbourg
  - Institut Gustave Roussy, Villejuif